CLINICAL TRIAL: NCT05289362
Title: Comparison of Efficacy of Basket and Balloon in the Removal of Pancreatic Duct Stones in Chronic Pancreatitis Under ERCP: a Single-blind, Parallel, Randomized Controlled Clinical Study
Brief Title: Comparison of Efficacy of Basket and Balloon in the Removal of Pancreatic Duct Stones in Chronic Pancreatitis Under ERCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH202202
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Pancreatitis, Chronic; Pancreatic Duct Stone
Keywords: Cholangiopancreatography, Endoscopic Retrograde
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treating pancreatic duct stones by using baskets (Experimental): ERCP will be performed under conscious sedation with intramuscular administration of diazepam 2.5-5.0 mg and pethidine 25-50 mg. If necessary, Endoscopic Sphincterotomy or Endoscopic Papillary Balloon Dilatation will be performed. A dilating bougie or balloon will be used to dilate the stenosis after sphincterotomy. After that, the basket will be used to remove the stones first, and the balloon will replace the basket after 15 minutes to remove any remaining stones. Finally, the effect of the basket will be evaluated.
  Interventions: Device: Basket group
- Treating pancreatic duct stones by using balloons (Active Comparator): ERCP will be performed under conscious sedation with intramuscular administration of diazepam 2.5-5.0 mg and pethidine 25-50 mg. If necessary, Endoscopic Sphincterotomy or Endoscopic Papillary Balloon Dilatation will be performed. A dilating bougie or balloon will be used to dilate the stenosis after sphincterotomy. After that, the balloon will be used to remove the stones first, and the basket will replace the balloon after 15 minutes to remove any remaining stones. Finally, the effect of the balloon will be evaluated.
  Interventions: Device: Balloon group

INTERVENTIONS:
Device: Basket group — Under ERCP, the basket is preferentially used to remove the pancreatic duct stones, and then the balloon is used to evaluate the effect and remove the residual stones.
  Arms: Treating pancreatic duct stones by using baskets
Device: Balloon group — Under ERCP, the balloon is preferentially used to remove the pancreatic duct stones, and then the basket is used to evaluate the effect and remove the residual stones.
  Arms: Treating pancreatic duct stones by using balloons

SUMMARY:
This study will compare the efficacy of basket and balloon in the removal of pancreatic duct stones under ERCP.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is an inflammatory disease that can causes progressive fibrosis of pancreatic tissue and eventually leads to damage of pancreatic exocrine and endocrine. According to statistics, the prevalence of CP in China is 13/10 million, which is still increasing. Pancreatic duct stones are the most important pathological changes of CP. More than 50% of patients with CP are accompanied by pancreatic duct stones, which can lead to pancreatic duct obstruction, hypertension and tissue ischemia. Removal of pancreatic duct stones under Endoscopic retrograde cholangiopancreatography (ERCP) are the first choice. ERCP is effective in the treatment of pancreatic duct stones (diameter < 5mm) located in the head/body of the pancreas by using basket and/or balloon catheter.

In the clinical work of investigators' center, the ERCP treatment of pancreatic duct stones also mainly adopts basket and balloon, but whether to try basket or balloon first is mainly determined by the subjective decision of the on-site endoscopist. More than 70% of patients use the above two tools in one ERCP operation, which aims to achieve better effect, but the order of the two tools is uncertain.

However, there is no relevant research on whether the first choice for the treatment of pancreatic duct stones is the basket or the balloon, or the combination of the two tools. This study will compare the efficacy of basket and balloon in the removal of pancreatic duct stones under ERCP, including the difference of stone clearance rate, abdominal pain score (Izbicki Pain Score), postoperative complications and medical expenses.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic adult patients diagnosed with chronic pancreatitis and pancreatic duct stones;
* stones (≤5 mm in diameter) are located in the main pancreatic duct of the pancreatic head/body with dilation of the proximal pancreatic duct.

Exclusion Criteria:

* suspected to have malignant tumors;
* history of pancreatic surgery or gastrojejunostomy (Billroth II);
* bile duct stricture secondary to cholangitis or chronic pancreatitis;
* acute pancreatitis exacerbation or acute exacerbation of chronic pancreatitis (including biliary pancreatitis);
* there is a stent in the main pancreatic duct;
* coagulation dysfunction (INR≥1.5 or platelet count≤50×10^9/L);
* pregnant or breastfeeding women;
* patients who refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-03-12 (Estimated)

PRIMARY OUTCOMES:
clearance rates of pancreatic duct stones | during ERCP procedure
  Clearance rates have been defined as complete, partial, or failure if the proportion of stones cleared was > 90%, 50% - 90%, or < 50%, respectively.

SECONDARY OUTCOMES:
timeout rate | during ERCP procedure
  Basket or balloon cannot completely remove stones in the targeted area of the pancreatic duct within 15 minutes.
time taken to completely clear the stone | during ERCP procedure
  The time taken by the basket or balloon to completely clear the stones in the targeted area of the pancreatic duct.
number of times to completely clear the stone | during ERCP procedure
  The number of attempts made by the basket or balloon to completely clear the stones in the targeted area of the pancreatic duct.
post-ERCP complications | 30 days after ERCP procedure
  Major post-ERCP complications includes post-ERCP pancreatitis, bleeding, infection, and perforation, which are classified as mild, moderate, or severe, depending mainly on the length of hospitalization and the need for invasive treatment.

OTHER OUTCOMES:
abdominal pain relief rate | 30 days after ERCP procedure
  Postoperative and preoperative abdominal pain was assessed using the Visual Analogue Scale (VAS). VAS can be calculated ranging from 0 (no pain) to 100 (severe pain).

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hao L, Liu Y, Xie T, Wang T, Guo HL, Pan J, Wang D, Bi YW, Ji JT, Xin L, Du TT, Lin JH, Zhang D, Zeng XP, Zou WB, Chen H, Li BR, Liao Z, Cong ZJ, Shi RH, Li ZS, Hu LH. Risk Factors and Nomogram for Pancreatic Stone Formation in Chronic Pancreatitis over a Long-Term Course: A Cohort of 2,153 Patients. Digestion. 2020;101(4):473-483. doi: 10.1159/000500941. Epub 2019 Jun 25. PMID 31238312
- [Background] Hu L, Sun X, Hao J, Xie T, Liu M, Xin L, Sun T, Liu M, Zou W, Ye B, Liu F, Wang D, Cao N, Liao Z, Li Z. Long-term follow-up of therapeutic ERCP in 78 patients aged 90 years or older. Sci Rep. 2014 May 13;4:4918. doi: 10.1038/srep04918. PMID 24819780